CLINICAL TRIAL: NCT06116669
Title: Effects of Oral Iron Supplementation Before vs at Time of Vaccination on Immune Response in Iron Deficient Kenyan Women
Acronym: DIVA_II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DIVA_II
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — COVID-19 Vaccines; Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-treatment group (Experimental): Participants assigned to this group will receive 100 mg oral iron daily on study days 1-56.
  Interventions: Dietary Supplement: Iron supplementation; Biological: MenACWY vaccine; Biological: COVID-19 vaccine; Biological: Typhim Vi vaccine
- Simultaneous treatment group (Experimental): Participants assigned to this group will receive placebo daily on study days 1-28 and 100 mg oral iron daily on study days 29-56.
  Interventions: Dietary Supplement: Iron supplementation; Biological: MenACWY vaccine; Biological: COVID-19 vaccine; Other: Placebo; Biological: Typhim Vi vaccine
- Control group (Placebo Comparator): Participants assigned to this group will receive placebo daily on study days 1-56.
  Interventions: Dietary Supplement: Iron supplementation; Biological: MenACWY vaccine; Biological: COVID-19 vaccine; Other: Placebo; Biological: Typhim Vi vaccine

INTERVENTIONS:
Dietary Supplement: Iron supplementation — Iron supplements as 100 mg oral iron as FeSO4 given daily
Biological: MenACWY vaccine — MenACWY vaccination given on day 28 to all participants
Biological: COVID-19 vaccine — Johnson & Johnson COVID- 19 (JJ COVID-19) vaccination given on day 28 to all participants
Other: Placebo — matching placebo capsules given daily
  Arms: Control group; Simultaneous treatment group
Biological: Typhim Vi vaccine — Typhim Vi vaccination given on day 28 to all participants

SUMMARY:
Iron deficiency (ID) anemia (IDA) is a global public health problem, with the highest prevalence in Africa. Vaccines often underperform in low- and middle-income countries (LMIC), and undernutrition, including ID, likely plays a role. Recent studies have shown the importance of iron status in vaccine response. Intravenous iron given at time of vaccination improved response to yellow fever and COVID-19 vaccines in IDA Kenyan women. Whether oral iron treatment would have a similar beneficial effect on vaccine response is uncertain. Also, timing of oral iron treatment needs further investigation.

The co-primary objectives of this study are to assess 1) whether IDA in Kenyan women impairs vaccine response, and whether oral iron treatment improves their response; 2) the timing of oral iron treatment to improve vaccine response (prior to vaccination vs at time of vaccination).

We will conduct a double-blind randomized controlled trial in southern Kenya to assess the effects of iron supplementation on response to three single-shot vaccines: Johnson & Johnson COVID- 19 (JJ COVID-19), the quadrivalent meningococcal vaccine (MenACWY) and the typhoid Vi polysaccharide vaccine (Typhim Vi). Women with IDA will be recruited and randomly assigned to three study groups: group 1 (pre- treatment) will receive 100 mg oral iron as ferrous sulfate (FeSO4) daily on days 1-56; group 2 (simultaneous treatment) will receive matching placebo daily on days 1-28, and 200 mg oral iron as FeSO4 daily on days 29-56; and group 3 (control) will receive matching placebo daily on days 1-56. Women in all groups will receive the JJ COVID-19 vaccine, the MenACWY and the Typhim Vi vaccine on day 28. Cellular immune response and serology will be measured at 28 days after vaccination in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial
* Female aged 18-49 years
* Moderate anemia (Hb <110 g/L, but not severely anemic with Hb <80 g/L)
* Iron deficient (ZnPP >40 mmol/mol haem)
* Anticipated residence in the study area for the study duration

Exclusion Criteria:

* Major chronic infecious disease (e.g., HIV infection);
* Major chronic non-infecious disease (e.g., Type 2 diabetes, cancer);
* Chronic medications;
* Use of iron-containing mineral and vitamin supplementation 2 weeks prior to study start;
* COVID-19 vaccine or confirmed COVID-19 infection within the past 2 years
* MenACWY vaccine in the past
* Typhim Vi vaccine in the past
* Pregnant (confirmed by rapid test during screening)
* Malaria (confirmed by rapid test) à study start will be postponed

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
JJ COVID-19 vaccine response | Day 56
  Anti-spike (S1) IgG and anti-receptor-binding domain (RBD) IgG against SARS-COV-2
MenACWY vaccine response | Day 56
  Measurement of antibody response against serogroups A, C, W, and Y.
Typhoid vaccine response | Day 56
  Measurement of antibody response against Typhoid

SECONDARY OUTCOMES:
Hemoglobin | Day 1
  iron status
Hemoglobin | Day 28
  iron status
Hemoglobin | Day 56
  iron status
Serum ferritin | Day 1
  iron status
Serum ferritin | Day 28
  iron status
Serum ferritin | Day 56
  iron status
soluble transferrin receptor | Day 1
  iron status
soluble transferrin receptor | Day 28
  iron status
soluble transferrin receptor | Day 56
  iron status
Plasma iron | Day 1
  iron status
Plasma iron | Day 28
  iron status
Plasma iron | Day 56
  iron status
Total iron binding capacity | Day 1
  iron status
Total iron binding capacity | Day 28
  iron status
Total iron binding capacity | Day 56
  iron status
Transferrin saturation | Day 1
  iron status
Transferrin saturation | Day 28
  iron status
Transferrin saturation | Day 56
  iron status
C- reactive protein | Day 1
  inflammation status
C- reactive protein | Day 28
  inflammation status
C- reactive protein | Day 56
  inflammation status
alpha- 1- glycoprotein | Day 1
  inflammation status
alpha- 1- glycoprotein | Day 28
  inflammation status
alpha- 1- glycoprotein | Day 56
  inflammation status
Retinol binding protein | Day 1
  Vitamin A status
Retinol binding protein | Day 28
  Vitamin A status
Retinol binding protein | Day 56
  Vitamin A status
Plasma zinc | Day 1
  Zinc status
COVID-19 specific T cell response | Day 28
  QuantiFERON SARS-CoV-2 whole blood assay - detection of IFN-gamma
COVID-19 specific T cell response | Day 56
  QuantiFERON SARS-CoV-2 whole blood assay - detection of IFN-gamma
COVID-19 specific T cell response | Day 28
  ELISpot assay on isolated peripheral blood mononuclear cells
COVID-19 specific T cell response | Day 56
  ELISpot assay on isolated peripheral blood mononuclear cells
Typhim Vi specific B-cell response | Day 28
  ELISpot assay on isolated peripheral blood mononuclear cells
Typhim Vi specific B-cell response | Day 56
  ELISpot assay on isolated peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Locations (1):
- Jomo Kenyatta University Of Agriculture And Technology, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No